CLINICAL TRIAL: NCT02762500
Title: A Randomized, Double-Blind, Placebo-Controlled Parallel Group Study to Assess the Efficacy and Safety of Induction Therapy With LYC-30937-EC in Subjects With Active Ulcerative Colitis
Brief Title: An Efficacy and Safety Study of LYC-30937-EC in Subjects With Active Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lycera Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LYC-30937-2001; 2016-000518-31 (EudraCT Number)
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Results first posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LYC-30937-EC 25 mg PO QD (Experimental): LYC-30937-EC 25 mg by mouth once daily for 8 weeks
  Interventions: Drug: LYC-30937-EC
- Placebo PO QD (Placebo Comparator): Matching placebo by mouth once daily for 8 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LYC-30937-EC
  Arms: LYC-30937-EC 25 mg PO QD
Drug: Placebo
  Arms: Placebo PO QD

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of LYC-30937-EC given orally once daily in subjects with active ulcerative colitis (UC) defined as a total Mayo score (TMS) of 4-11 inclusive, with an endoscopic score of ≥ 2 and a rectal bleeding score of ≥ 1 at screening.

DETAILED DESCRIPTION:
Approximately 120 subjects will be randomized to receive either enteric-coated (EC) LYC-30937-EC 25 mg PO once daily (QD) or matching placebo PO QD for the duration of 8 weeks. Randomization will be stratified based on previous exposure to anti-tumor necrosis factor (TNF) agents such that at least 50% of the randomized subjects will be anti-TNF naïve .

The study will consist of 3 phases:

* screening phase: up to 4 weeks
* double-blind placebo-controlled phase treatment: 8 weeks
* post-treatment follow-up: 2 weeks

Eligible subjects will be randomized at Week 0 (Study Day 1) to either LYC-30937-EC 25 mg or placebo. Screening will occur from Study Days -28 to -1. Randomization and first dosing will occur at Week 0/Study Day 1. Double-blind study visits will occur at Weeks 2, 4, and 8, with the last dose at Week 8/Study Day 57. Subjects will return at Week 10 for a post-treatment safety follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Clinical UC diagnosis ≥ 6 months prior to screening with minimum disease extent of ≥ 15cm from anal verge.
* Active UC defined as a TMS of 4-11 (inclusive) with endoscopic subscore of ≥ 2 and rectal bleeding subscore of ≥ 1 at screening.
* Females of childbearing potential must have a negative pregnancy test at screening and baseline visits and must agree to use acceptable methods of birth control while in the trial and for 30 days after taking the last dose of study drug.
* May be currently receiving treatment with oral aminosalicylates (ASA) for ≥ 6 weeks at a stable dose for ≥ 3 weeks prior to the screening screening endoscopy and/or thiopurine at a stable dose ≥ 8 weeks prior to the screening endoscopy and/or prednisone (dose 20 mg daily) or equivalent for ≥ 4 weeks and receiving stable dose for ≥ 2 weeks prior to screening endoscopy
* able to provide written informed consent and be compliant with study procedures.

Exclusion Criteria:

* History of Crohn's disease (CD) or indeterminate colitis or the presence or history of fistula consistent with CD.
* Presence of colon polyps.
* Severe extensive disease that in the investigators discretion is likely to require colonic surgery during the 8 week double-blind portion of the trial (eg, fulminant colitis, toxic megacolon, bowel perforation, evidence of acute abdomen).
* History of alcohol or drug abuse within 1 year of randomization.
* History of cancer including solid tumors and hematological malignancies (except basal cell and in situ squamous cell carcinomas of the skin that have been adequately treated with no recurrence for ≥ 1 year prior to screening.
* History or currently active primary or secondary immunodeficiency.
* Clinically relevant hepatic, neurologic, pulmonary, ophthalmological, gastrointestinal, endocrine, psychiatric, or other major systemic disease making implementation of the study difficult or that would put the subject at risk by participating in the study
* Positive test for Clostridium difficile or positive stool culture for enteric pathogens or presence of ova or parasites at screening.
* Liver function tests > 1.5 x upper limit of normal (ULN) or direct bilirubin > 1.5 x ULN
* Hemoglobin < 8.5 g/dl
* Neutrophils < 1500/mm3
* White blood cell (WBC) count < 3000/mm3
* Platelets < 80000 mm3
* International normalized ratio (INR) > 1.5
* Treatment with an immunosuppressant agent within 8 weeks of screening.
* Previous exposure to ≥ 2 approved or investigational biologic agents to treat UC.
* History of UC treatment with a biologic agent within 12 weeks of screening.
* Treatment with rectal steroids within 2 weeks of screening.
* Treatment with an investigational agent within 30 days of screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2016-07; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Jeffrey Wilkins, MD, Study Director — Lycera Corp.
Locations (58):
- United States (25):
  - Lycera Investigational Site, Little Rock, Arkansas
  - Lycera Investigational Site, Long Beach, California
  - Lycera Investigational Site, Mission Hills, California
  - Lycera Investigational Site, Rialto, California
  - Lycera Investigational Site, Hollywood, Florida
  - Lycera Investigational Site, Miami, Florida
  - Lycera Investigational Site, Decatur, Georgia
  - Lycera Investigational Site, Marietta, Georgia
  - Lycera Investigational Site, Chicago, Illinois
  - Lycera Investigational Site, Louisville, Kentucky
  - Lycera Investigational Site, Baton Rouge, Louisiana
  - Lycera Investigational Site, Ann Arbor, Michigan
  - Lycera Investigational Site, Brooklyn, New York
  - Lycera Investigational Site, New York, New York
  - Lycera Investigational Site, The Bronx, New York
  - Lycera Investigational Site, Greenville, North Carolina
  - Lycera Investigational Site, Flourtown, Pennsylvania
  - Lycera Investigational Site, Philadelphia, Pennsylvania
  - Lycera Investigational Site, Sayre, Pennsylvania
  - Lycera Investigational Site, Nashville, Tennessee
  - Lycera Investigational Site, Union City, Tennessee
  - Lycera Investigational Site., Houston, Texas
  - Lycera Investigational Sites, Houston, Texas
  - Lycera Investigational Site, Houston, Texas
  - Lycera Investigational Site, San Antonio, Texas
- Canada (2):
  - Lycera Investigational Site, Victoria, British Columbia
  - Lycera Investigational Site, Toronto, Ontario
- Czechia (4):
  - Lycera Investigational Site, Ostrava
  - Lycera Investigational Site, Prague
  - Lycera Investigational Site, Slaný
  - Lycera Investigational Site, Ústí nad Labem
- Hungary (3):
  - Lycera Investigational Site, Budapest
  - Lycera Investigational Site, Debrecen
  - Lycera Investigational Site, Hatvan
- Netherlands (2):
  - Lycera Investigational Site, Amsterdam
  - Lycera Investigational Site, Rotterdam
- Poland (17):
  - Lycera Investigational Site, Bydgoszcz
  - Lycera Investigational Site, Katowice
  - Lycera Investigational Site, Kielce
  - Lycera Investigational Site, Krakow
  - Lycera Investigational Site, Ksawerów
  - Lycera Investigational Site, Lodz
  - Lycera Investigational Site, Lublin
  - Lycera Investigational Site, Nowa Sól
  - Lycera Investigational Site, Piaseczno
  - Lycera Investigational Site, Poznan
  - Lycera Investigational Site, Skierniewice
  - Lycera Investigational Site, Sopot
  - Lycera Investigational Site, Staszów
  - Lycera Investigational Site, Szczecin
  - Lycera Investigational Site, Warsaw
  - Lycera Investigational Site, Wroclaw
  - Lycera Investigational Site, Włocławek
- Serbia (5):
  - Lycera Investigational Site, Belgrade
  - Lycera Investigational Site, Kragujevac
  - Lycera Investigational Site, Niš
  - Lycera Investigational Site, Subotica
  - Lycera Investigational Site, Zrenjanin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 42 study centers within the United States, Poland, Hungary, Czech Republic, Serbia and Netherlands. Study centers included academic medical centers and non-academic medical clinics.
Pre-assignment Details: Participants were 18 to 75 years of age with active ulcerative colitis for at least 6 months prior to screening, had a total Mayo score (TMS) ≥ 4 to ≤ 11, with endoscopic subscore ≥ 2, and rectal bleeding subscore ≥ 1 at screening.
Groups:
- LYC-30937-EC: LYC-30937-EC 25 mg by mouth once daily for 8 weeks
- Placebo: Matching placebo by mouth once daily for 8 weeks
Period: Overall Study
Arm/Group | LYC-30937-EC | Placebo
Started | 62 | 62
Completed | 60 | 59
Not Completed | 2 | 3
Not completed — Lack of Efficacy | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LYC-30937-EC | Placebo | Total
Number analyzed (Participants) | 62 | 62 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (11.94) | 39.3 (13.26) | 41.5 (12.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 25 | 52
  Male | 35 | 37 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 59 | 58 | 117
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 1 | 2 | 3
  White | 60 | 59 | 119
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 2 | 1 | 3
  Hungary | 1 | 1 | 2
  United States | 11 | 17 | 28
  Czechia | 3 | 2 | 5
  Poland | 43 | 38 | 81
  Serbia | 2 | 3 | 5
Baseline Total Mayo Score (TMS) and Modified Mayo Score (MMS) [Mean (Standard Deviation); unit: units on a scale] — TMS range: 0 (normal/no disease) to 12 (severe disease). TMS comprised of 4 subscores: stool frequency subscore, rectal bleeding subscore, endoscopy subscore, physician's global assessment subscore.
  MMS range: 0 (normal/no disease) to 9 (severe disease). MMS comprised of 3 subscores: stool frequency subscore, rectal bleeding subscore, endoscopy subscore. Population: One subject in the placebo treatment arm did not have a complete Mayo score at baseline and therefore they were not included in this analysis population.
  units on a scale
    Baseline TMS Mean (Standard Deviation): number analyzed (Participants) | 62 | 61 | 123
    Baseline TMS Mean (Standard Deviation) | 7.9 (1.46) | 7.8 (1.77) | 7.9 (1.62)
    Baseline MMS Mean (Standard Deviation) | 6.0 (1.38) | 5.7 (1.55) | 5.8 (1.47)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Achieve Clinical Remission at Week 8 Using Modified Mayo Score.
Description: The modified Mayo score is a tool designed to measure disease activity for ulcerative colitis. Scoring ranges from 0 to 9 points and consists of 3 subscores (stool frequency, rectal bleeding, endoscopy), each graded 0 to 3 with higher score indicating more severe disease activity. Endoscopy scoring was performed centrally.
  Clinical remission on the modified Mayo score was defined as a Mayo stool frequency subscore of ≤ 1, Mayo rectal bleeding subscore of 0 and a Mayo endoscopy subscore of ≤ 1.
Time Frame: 8 weeks
Population: The analysis population consisted of all randomized subjects (Full Analysis Set).
Measure: Count of Participants; unit: Participants
Groups:
- LYC-30937-EC 25 mg PO QD: LYC-30937-EC 25 mg by mouth once daily for 8 weeks
  LYC-30937-EC
- Placebo PO QD: Matching placebo by mouth once daily for 8 weeks
  Placebo
Arm/Group | LYC-30937-EC 25 mg PO QD | Placebo PO QD
Number analyzed (Participants) | 62 | 62
Participants | 7 | 12
Statistical Analysis 1: Comparison: LYC-30937-EC 25 mg PO QD vs Placebo PO QD; The response rate difference is the mean difference in response rates between the treatment and placebo responders. The p-value is based on one-sided Pearson chi-square test; Test type: Superiority; p = 0.106, Chi-squared — one-sided p-value; Statistical test was a one-sided performed at the 5% level of significance. Pearson chi-square test was used to test the null hypothesis; Risk Difference (RD) = -8.1, 90% CI 2-sided [-18.6 to 2.5] — 90% CI obtained based on normal approximation

2. Secondary Outcome: Number of Subjects Who Achieve Clinical Remission at Week 8 Using the Total Mayo Score.
Description: The total Mayo score is a tool designed to measure disease activity for ulcerative colitis. Scoring ranges from 0 to 12 points and consists of 4 subscores (stool frequency, rectal bleeding, endoscopy, physicians global assessment), each graded 0 to 3 with higher score indicating more severe disease activity. Endoscopy scoring was performed centrally.
  Clinical remission on the total Mayo Score is defined as a total Mayo score of ≤ 2, with no individual subscore > 1.
Time Frame: 8 weeks
Population: The analysis population consisted of all randomized subjects (Full Analysis Set).
Measure: Count of Participants; unit: Participants
Arm/Group | LYC-30937-EC 25 mg PO QD | Placebo PO QD
Number analyzed (Participants) | 62 | 62
Participants | 7 | 12
Statistical Analysis 1: Comparison: LYC-30937-EC 25 mg PO QD vs Placebo PO QD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.106, Chi-squared — one-sided p-value; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = -8.1, 90% CI 2-sided [-18.6 to 2.5] — 90% CI obtained based on normal approximation

3. Secondary Outcome: Number of Subjects With a Clinical Response on the Modified Mayo Score at Week 8.
Description: The modified Mayo score is a tool designed to measure disease activity for ulcerative colitis. Scoring ranges from 0 to 9 points and consists of 3 subscores (stool frequency, rectal bleeding, endoscopy), each graded 0 to 3 with higher score indicating more severe disease activity. Endoscopy scoring was performed centrally.
  Clinical response on the modified Mayo score at Week 8 was defined as a reduction from the baseline modified Mayo score of ≥ 2 points and ≥ 25%, and a decrease from baseline in rectal bleeding score of ≥ 1 point or absolute rectal bleeding score of ≤ 1 point.
Time Frame: 8 weeks
Population: The analysis population consisted of all randomized subjects (Full Analysis Set).
Measure: Count of Participants; unit: Participants
Arm/Group | LYC-30937-EC 25 mg PO QD | Placebo PO QD
Number analyzed (Participants) | 62 | 62
Participants | 32 | 36
Statistical Analysis 1: Comparison: LYC-30937-EC 25 mg PO QD vs Placebo PO QD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.235, Chi-squared — one-sided p-value; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = -6.5, 90% CI 2-sided [-21.1 to 8.2] — 90% CI obtained based on normal approximation

4. Secondary Outcome: Number of Subjects With a Clinical Response on the Total Mayo Score at Week 8.
Description: The total Mayo score is a tool designed to measure disease activity for ulcerative colitis. Scoring ranges from 0 to 12 points and consists of 4 subscores (stool frequency, rectal bleeding, endoscopy, physicians global assessment), each graded 0 to 3 with higher score indicating more severe disease activity. Endoscopy scoring was performed centrally.
  Clinical response on the total Mayo score at Week 8 was defined as a reduction from baseline total Mayo score of ≥ 3 points and ≥ 30%, and a decrease from baseline in rectal bleeding score of ≥ 1 point or absolute rectal bleeding score of ≤ 1 point.
Time Frame: 8 weeks
Population: The analysis population consisted of all randomized subjects (Full Analysis Set).
Measure: Count of Participants; unit: Participants
Arm/Group | LYC-30937-EC 25 mg PO QD | Placebo PO QD
Number analyzed (Participants) | 62 | 62
Participants | 26 | 32
Statistical Analysis 1: Comparison: LYC-30937-EC 25 mg PO QD vs Placebo PO QD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.140, Chi-squared — one-sided p-value; [statistical method as in outcome 1, analysis 1]; Risk Difference (RD) = -9.7, 90% CI 2-sided [-24.3 to 5.0] — 90% CI obtained based on normal approximation

5. Secondary Outcome: Percent Change From Baseline to Week 8 in Fecal Calprotectin in Subjects With Baseline Fecal Calprotectin ≥ 250 µg/g
Description: Fecal calprotectin is an indicator of inflammation in the colon with higher levels indicative of higher levels of inflammation.
Time Frame: Baseline to Week 8
Population: All randomized subjects who had an elevated baseline fecal calprotectin level of ≥ 250 µg/g and who had both a baseline and Week 8 value.
Measure: Least Squares Mean (Standard Error); unit: percent change from baseline
Arm/Group | LYC-30937-EC 25 mg PO QD | Placebo PO QD
Number analyzed (Participants) | 51 | 44
percent change from baseline | -35.22 (13.81) | 9.37 (15.07)
Statistical Analysis 1: Comparison: LYC-30937-EC 25 mg PO QD vs Placebo PO QD; Subjects included in this analysis were those with a baseline fecal calprotectin value ≥ 250 µg/g; Test type: Superiority; p = 0.032, ANCOVA; The mean change from baseline at Week 8 was analyzed using ANCOVA with a factor for treatment and a covariate for baseline scores; Mean Difference (Final Values) = -44.59, 90% CI 2-sided [-78.66 to -10.53]

6. Secondary Outcome: Percent Change From Baseline in Total Mayo Score at Week 8.
Description: Analyzes the change in total Mayo score score between baseline and Week 8 for all randomized subjects who had total Mayo score scores at both baseline and Week 8.
  The total Mayo score is a tool designed to measure disease activity for ulcerative colitis. Scoring ranges from 0 to 12 points and consists of 4 subscores (stool frequency, rectal bleeding, endoscopy, physicians global assessment), each graded 0 to 3 with higher score indicating more severe disease activity. Endoscopy scoring was performed centrally.
Time Frame: Baseline to Week 8
Population: All randomized subjects randomized who had TMS scores at baseline and Week 8.
Measure: Least Squares Mean (Standard Error); unit: Percent Change from baseline
Arm/Group | LYC-30937-EC 25 mg PO QD | Placebo PO QD
Number analyzed (Participants) | 59 | 58
Percent Change from baseline | -2.49 (0.33) | -2.67 (0.33)
Statistical Analysis 1: Comparison: LYC-30937-EC 25 mg PO QD vs Placebo PO QD; Test type: Superiority; p = 0.708, ANCOVA; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = 0.18, 90% CI 2-sided [-0.60 to 0.95]

7. Other Pre Specified Outcome: Number of Subjects With Type of Adverse Events (AEs) Serious Adverse Events (SAEs) and AEs That Led to Discontinuation of Treatment.
Description: Adverse events (AEs) were collected from the time a subject signed the informed consent. Treatment-emergent adverse events (TEAEs) are AEs occurring or worsening after the first dose of study drug (LYC-30937-EC 25 mg or placebo). Adverse event severity was assessed by the Investigator using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v 4.03, with grading as follows: Grade 1 = mild (asymptomatic or mild symptoms), Grade 2 = moderate (minimal, local intervention, or noninvasive intervention indicated); Grade 3 = severe (or medically significant but not life-threatening); Grade 4 = life-threatening; Grade 5 = death.
Time Frame: 10 weeks
Population: Safety Set, consisting of all randomized subjects who took at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | LYC-30937-EC 25 mg PO QD | Placebo PO QD
Number analyzed (Participants) | 62 | 62
Participants
  Subjects with ≥ 1 TEAE | 22 | 27
  Subjects with ≥ 1 TESAE | 1 | 3
  Subjects with TEAE leading to discontinuation | 0 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time a subject signed informed consent through the Week 10 follow-up visit. SAEs occurring after the last study visit that were determined by the investigator to be related to study drug were to be reported.
Arm/Group | LYC-30937-EC 25 mg PO QD | Placebo PO QD
All-Cause Mortality (participants affected / at risk) | 0/62 | 0/62
Serious Adverse Events (participants affected / at risk) | 1/62 | 3/62
Other Adverse Events (participants affected / at risk) | 10/62 | 11/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LYC-30937-EC 25 mg PO QD (N=62) | Placebo PO QD (N=62)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LYC-30937-EC 25 mg PO QD (N=62) | Placebo PO QD (N=62)
Headache (Nervous system disorders) | 6 (6) | 5 (6)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 6 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Center results cannot be submitted for publication before results of multicenter study are published unless it is more than 1 year since study completion. Then Investigator can publish if manuscript is submitted to Lycera ≥ 60 days prior to submission (or per Investigator contract). If Lycera decides publication would hinder development, Investigator must delay submission. Investigator must delete confidential information before submission and defer publication to allow patent applications.

DOCUMENTS (2):
  • Study Protocol (2017-06-05): https://cdn.clinicaltrials.gov/large-docs/00/NCT02762500/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT02762500/SAP_001.pdf